CLINICAL TRIAL: NCT04456530
Title: Use of Testosterone to Prevent Post-Surgical Muscle Loss - Pilot Study
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The Stone Research Foundation for Sports Medicine and Arthritis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SRF-030
Record Dates: First submitted 2020-06-24; First posted 2020-07-02 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Muscle Atrophy; Surgery; Knee Injuries and Disorders; Complication of Surgical Procedure; Trauma
Keywords: Surgery; Testosterone; Muscle atrophy; Post-operative rehabilitation
MeSH Terms: conditions — Muscular Atrophy; Knee Injuries; Disease; Wounds and Injuries | interventions — Testosterone Propionate; Injections, Intramuscular; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Both the participant and analyzing MRI Radiologist will be blind.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Testosterone Group (Experimental): Participants receiving two IM Testosterone injections.
  Interventions: Drug: Aveed 750 MG in 3 ML IM Injection
- Control Group (Placebo Comparator): Participants receiving two IM Normal Saline Injections.
  Interventions: Other: Normal Saline 3 ML IM Injection

INTERVENTIONS:
Drug: Aveed 750 MG in 3 ML IM Injection — Participants in the Testosterone Group will receive two IM Aveed injections 1 month apart.
  Arms: Testosterone Group
Other: Normal Saline 3 ML IM Injection — Participants in the Control Group will receive two IM normal saline injections 1 month apart.
  Arms: Control Group

SUMMARY:
The loss of muscle mass post-surgery confounds recovery efforts and leads to a delay in patient's ability to return to activities. Although the use of testosterone in aging and chronic muscle loss has been investigated, this study could prove short-term use of testosterone efficacious in preventing muscle atrophy due to surgery. We hypothesize that by bracketing an indexed knee surgery with testosterone undecanoate injections, post-surgical quadriceps muscle loss may be minimized. Determination of the effect of intra-muscular (IM) testosterone injections in preventing quadriceps muscle loss are measured by serial MRI and manual measurements of quadriceps cross-section.

DETAILED DESCRIPTION:
This is an in vivo study using serial IM testosterone undeconate injections in participants undergoing knee surgery with limited weight bearing post-operatively which includes partial/total knee replacement, ACL reconstruction/revision, meniscal allograft transplantation and articular cartilage paste grafting. The design is a randomized, controlled, double blind, longitudinal study of intra-muscular injections of testosterone versus saline control. Pre-operative and post-operative assessments will include: serial MRIs and manual measurements of quadriceps cross-section and knee pain and function survey, KOOS. Blood analysis will be performed for therapeutic assessment and safety. The participant will receive two testosterone undeconate injections, once during their pre-operative visit and once during their 1 month visit. Timing of assessments will be pre-operative, 1-4 days post-operative and 1, 3, and 6 months. Measurement of the control group versus experimental group at all time points may identify differences in participant response to testosterone injections.

ELIGIBILITY:
Inclusion Criteria:

* Males age 18-65.
* Undergoing significant knee surgery such as partial/total knee replacement, ligament reconstruction, meniscus surgeries or articular cartilage paste grafting.

Exclusion Criteria:

* Men with carcinoma of the breast or known or suspected carcinoma of the prostate.
* Men with BMI > 30 and Type I or II diabetes diagnosis
* Men prone to deep vein thrombosis or sleep apnea.
* Men with pre-existing hematocrit abnormalities.
* Men with pre-existing cardiac, renal, hepatic disease.
* Men who are taking insulin, medicines that decrease blood clotting or corticosteroids.
* Men with known hypersensitivity to testosterone undecanoate or any of its formulation ingredients (testosterone, refined castor oil, benzyl benzoate).
* Subject's unable or unwilling to comply with the protocol.
* Subject's unable to provide informed consent.
* Subject's unable to understand verbal and/or written English.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-05-08 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in MRI Cross Sectional Area of the Quadriceps | Pre-operative and 1, 3, and 6 months post-operative
  T1 Axial and Sagittal planes will be obtained using a ONI 1.0T extremity MRI. Axial Cross sectional Area (cm^2) will be measured of the Quadriceps muscle.
Change in Manual Measurements of the Quadriceps | Pre-operative and 1, 3, and 6 months post-operative
  Manual measurement of the quadriceps muscle will be performed 8-cm proximal to the superior-patella using a standard cm measuring tape.

SECONDARY OUTCOMES:
Change in Knee Pain and Function Survey, KOOS | Pre-operative and 1, 3, and 6 months post-operative
  Evaluate the knee pain and function of subjects as measures by the KOOS assessment.
  Sections:
  1. Pain
  2. Symptoms
  3. Activities of Daily Living
  4. Sports and Recreation
  5. Quality of Life
  Scoring:
  Each subscale score is calculated independently. The mean score of the individual items of each subscale is calculated and divided by 4 (the highest possible score for a single answer option). Traditionally in orthopedics, 100 indicates no problems and 0 indicates extreme problems. The normalized score is transformed to meet this standard.

OTHER OUTCOMES:
Change in serum cortisol (mcg/dL) levels | Pre-operative, 1-4 days post-operative and 1 month and 3 months post-operative
  Laboratory blood analysis of cortisol will be performed for therapeutic assessment and safety.
Change in serum testosterone (ng/dL) levels | Pre-operative, 1-4 days post-operative and 1 month and 3 months post-operative
  Laboratory blood analysis of testosterone will be performed for therapeutic assessment and safety.
Change in serum prostate specific antigen (ng/mL) levels | Pre-operative, 1-4 days post-operative and 1 month and 3 months post-operative
  Laboratory blood analysis of PSA will be performed for therapeutic assessment and safety.
Change in serum hepatic function panel (mg/dL) levels | Pre-operative, 1-4 days post-operative and 1 month and 3 months post-operative
  Laboratory blood analysis of HFP will be performed for therapeutic assessment and safety.
Change in complete blood count with differential levels | Pre-operative, 1-4 days post-operative and 1 month and 3 months post-operative
  Laboratory blood analysis CBC w/ diff will be performed for therapeutic assessment and safety.

CONTACTS AND LOCATIONS:
Overall Officials: Mani Vessal, Ph.D., Study Director — Stone Research Foundation
Locations (1):
- Stone Research Foundation, San Francisco, California, United States

REFERENCES:
- [Background] Bassil N, Alkaade S, Morley JE. The benefits and risks of testosterone replacement therapy: a review. Ther Clin Risk Manag. 2009 Jun;5(3):427-48. doi: 10.2147/tcrm.s3025. Epub 2009 Jun 22. PMID 19707253
- [Background] Nicholas JJ, Taylor FH, Buckingham RB, Ottonello D. Measurement of circumference of the knee with ordinary tape measure. Ann Rheum Dis. 1976 Jun;35(3):282-4. doi: 10.1136/ard.35.3.282. PMID 984911
- [Background] Arangio GA, Chen C, Kalady M, Reed JF 3rd. Thigh muscle size and strength after anterior cruciate ligament reconstruction and rehabilitation. J Orthop Sports Phys Ther. 1997 Nov;26(5):238-43. doi: 10.2519/jospt.1997.26.5.238. PMID 9353686
- [Background] Marcon M, Ciritsis B, Laux C, Nanz D, Nguyen-Kim TD, Fischer MA, Andreisek G, Ulbrich EJ. Cross-sectional area measurements versus volumetric assessment of the quadriceps femoris muscle in patients with anterior cruciate ligament reconstructions. Eur Radiol. 2015 Feb;25(2):290-8. doi: 10.1007/s00330-014-3424-2. Epub 2014 Oct 31. PMID 25358592
- [Background] Ruhdorfer AS, Dannhauer T, Wirth W, Cotofana S, Roemer F, Nevitt M, Eckstein F; OAI investigators. Thigh muscle cross-sectional areas and strength in knees with early vs knees without radiographic knee osteoarthritis: a between-knee, within-person comparison. Osteoarthritis Cartilage. 2014 Oct;22(10):1634-8. doi: 10.1016/j.joca.2014.06.002. PMID 25278072
- [Background] Orgiu S, Lafortuna CL, Rastelli F, Cadioli M, Falini A, Rizzo G. Automatic muscle and fat segmentation in the thigh from T1-Weighted MRI. J Magn Reson Imaging. 2016 Mar;43(3):601-10. doi: 10.1002/jmri.25031. Epub 2015 Aug 13. PMID 26268693
- [Background] Hartgens F, Kuipers H. Effects of androgenic-anabolic steroids in athletes. Sports Med. 2004;34(8):513-54. doi: 10.2165/00007256-200434080-00003. PMID 15248788
- [Background] Irrgang JJ, Ho H, Harner CD, Fu FH. Use of the International Knee Documentation Committee guidelines to assess outcome following anterior cruciate ligament reconstruction. Knee Surg Sports Traumatol Arthrosc. 1998;6(2):107-14. doi: 10.1007/s001670050082. PMID 9604196
- [Background] Brazier JE, Harper R, Jones NM, O'Cathain A, Thomas KJ, Usherwood T, Westlake L. Validating the SF-36 health survey questionnaire: new outcome measure for primary care. BMJ. 1992 Jul 18;305(6846):160-4. doi: 10.1136/bmj.305.6846.160. PMID 1285753
- [Background] Amory JK, Chansky HA, Chansky KL, Camuso MR, Hoey CT, Anawalt BD, Matsumoto AM, Bremner WJ. Preoperative supraphysiological testosterone in older men undergoing knee replacement surgery. J Am Geriatr Soc. 2002 Oct;50(10):1698-701. doi: 10.1046/j.1532-5415.2002.50462.x. PMID 12366624
- [Background] Griggs RC, Kingston W, Jozefowicz RF, Herr BE, Forbes G, Halliday D. Effect of testosterone on muscle mass and muscle protein synthesis. J Appl Physiol (1985). 1989 Jan;66(1):498-503. doi: 10.1152/jappl.1989.66.1.498. PMID 2917954
- [Background] Akima H, Furukawa T. Atrophy of thigh muscles after meniscal lesions and arthroscopic partial menisectomy. Knee Surg Sports Traumatol Arthrosc. 2005 Nov;13(8):632-7. doi: 10.1007/s00167-004-0602-9. Epub 2005 Apr 13. PMID 15827765
- [Background] Wu B, Lorezanza D, Badash I, Berger M, Lane C, Sum JC, Hatch GF 3rd, Schroeder ET. Perioperative Testosterone Supplementation Increases Lean Mass in Healthy Men Undergoing Anterior Cruciate Ligament Reconstruction: A Randomized Controlled Trial. Orthop J Sports Med. 2017 Aug 9;5(8):2325967117722794. doi: 10.1177/2325967117722794. eCollection 2017 Aug. PMID 28840147